CLINICAL TRIAL: NCT04243369
Title: Collaboration Live Clinical Study
Brief Title: Collaboration Live
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philips Clinical & Medical Affairs Global (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: US-GIS-10649
Record Dates: First submitted 2020-01-21; First posted 2020-01-28 (Actual); Results first posted 2020-12-04 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-11

CONDITIONS: Pregnancy Related
Keywords: Collaboration Live; Telemedicine; Ultrasound

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Experimental - Collaboration Live software (Other)
  Interventions: Device: Non-diagnostic software solution

INTERVENTIONS:
Device: Non-diagnostic software solution — Collaboration Live is a non-diagnostic software solution intended for use with Philips (Philips Ultrasound, 22100 Bothell Everett Highway, Bothell, Washington 98021) EPIQ and Affiniti Series Ultrasound Systems (software version 5.0.2) that allows users to communicate (by text, voice, screen share, webcam video and remote takeover) from an ultrasound system or workstation to a remote destination.

SUMMARY:
Collaboration Live is a prospective, single-arm clinical study of subjects who provide written consent. Subjects are scanned using a Philips EPIQ 5 or EPIQ 7 Ultrasound System equipped with Collaboration Live software. The study investigator will evaluate performance of the Collaboration Live tool with regard to performance of conferencing, sharing and control capabilities. Adverse events will be reported and the study investigator will assess potential relationship to the study device or study procedure. Additionally, the utility of Collaboration Live in remote consult of study patients will be evaluated. No patient follow-up beyond the initial consultation will be conducted with the Collaboration Live software solution.

ELIGIBILITY:
Inclusion Criteria:

* Subject is at least 18 years of age
* Subject in indicated for a routine Obstetrics/Gynecology ultrasound examination at the site.
* Subject is willing and capable of providing informed consent and participating in this study

Exclusion Criteria:

* A medical condition or co-morbidity that would be unduly affected by study participation, per investigator discretion

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Subject in indicated for a routine OB/GYN ultrasound examination at the site.
Enrollment: 30 (Actual)
Dates: Start 2020-01-09 (Actual); Primary Completion 2020-02-20 (Actual); Study Completion 2020-02-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Perinatal Associates of New Mexico, Albuquerque, New Mexico
  - Perinatal Associates of New Mexico, Rio Rancho, New Mexico
  - Perinatal Associates of New Mexico, Santa Fe, New Mexico

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Experimental - Collaboration Live Software
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Experimental - Collaboration Live Software
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.6 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 30
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 30
Gestational age [Mean (Standard Deviation); unit: weeks] | 27.8 (6.6)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 34.0 (7.0)

OUTCOME MEASURES:

1. Primary Outcome: Rate of Clinically Acceptable Performance of Remote Control Functionality
Description: The system responds to the remote input as intended and without a delay interfering with the conduct of the exam. Additionally, a clinically acceptable exam would result in no adverse events related to the control feature
Time Frame: Intra-procedural (1 day)
Measure: Number (95% Confidence Interval); unit: Percentage of total exams
Arm/Group | Experimental - Collaboration Live Software
Number analyzed (Participants) | 30
Percentage of total exams | 100 [88.4 to 100]
Statistical Analysis 1: Comparison: Experimental - Collaboration Live Software; Test type: Other — Only descriptive statistics was provided. The rate and the exact 95% CI of the rate using the Clopper-Pearson Exact method is calculated; Rate = 100, 95% CI 2-sided [88.4 to 100]

2. Secondary Outcome: Number of Participants With Technical Issues
Description: Number of subjects for which device deficiencies are reported
Time Frame: Intra-procedural (1 day)
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental - Collaboration Live Software
Number analyzed (Participants) | 30
Participants | 2

3. Secondary Outcome: Success Rates for Key Tasks in the Collaborative Exam
Description: Establishing the remote connection, establishing text chat, establishing voice call, establishing webcam feed, establishing screen share, establishing remote control
Time Frame: Intra-procedural (1 day)
Measure: Number; unit: percentage of participants
Arm/Group | Experimental - Collaboration Live Software
Number analyzed (Participants) | 30
percentage of participants | 100

4. Secondary Outcome: Travel Reduction Attributable to Use of Collaboration Live
Description: Distance between the scanning facility and the investigator's location will be recorded (in miles).
Time Frame: Intra-procedural (1 day)
Measure: Mean (Standard Deviation); unit: miles
Arm/Group | Experimental - Collaboration Live Software
Number analyzed (Participants) | 30
miles | 38.0 (18.6)

5. Secondary Outcome: Ease of Use
Description: 5-point (Likert) scale data will be reported by the investigator.( 5 = Strongly agree, 4 = Agree, 3 = Neutral, 2 = Disagree, 1 = Strongly disagree)
Time Frame: Intra-procedural (1 day)
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental - Collaboration Live Software
Number analyzed (Participants) | 30
Participants
  Physician assessment: Strongly Agree | 26
  Physician assessment: Agree | 4
  Sonographer Assessment: Strongly Agree | 28
  Sonographer Assessment: Agree | 2

6. Secondary Outcome: User Feedback Regarding Streaming, Image Quality and Overall Experience
Description: 5-point (Likert) scale data will be reported by the investigator. ( 5 = Very good, 4 = Good, 3 = Acceptable, 2 = Poor, 1 = Very Poor)
Time Frame: Intra-procedural (1 day)
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental - Collaboration Live Software
Number analyzed (Participants) | 30
Participants
  Physician Assessment: Acceptable | 0
  Physician Assessment: Good | 3
  Physician Assessment: Very Good | 27
  Sonorapher: Acceptable | 1
  Sonorapher: Good | 4
  Sonorapher: Very Good | 25

7. Secondary Outcome: Patient Feedback Regarding Remote Consultation
Description: Tele-medicine Satisfaction Questionnaire
Time Frame: 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental - Collaboration Live Software
Number analyzed (Participants) | 30
Participants
  Good | 0
  Very Good | 30

8. Secondary Outcome: Impact of Remote Consultation on Reimbursement
Description: Submitted charges and reimbursement rates for remote patient consultation data will be recorded and compared to standard rates for in-person consultation
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: percentage of standard amount
Arm/Group | Experimental - Collaboration Live Software
Number analyzed (Participants) | 30
percentage of standard amount | 96.9 (7.2)

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | Experimental - Collaboration Live Software
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Statistical Analysis Plan (2020-01-16): https://cdn.clinicaltrials.gov/large-docs/69/NCT04243369/SAP_000.pdf
  • Study Protocol (2019-10-24): https://cdn.clinicaltrials.gov/large-docs/69/NCT04243369/Prot_001.pdf